CLINICAL TRIAL: NCT06041620
Title: A Study to Evaluate the Efficacy and Safety of Autologous CRISPR-Cas12b Edited Hematopoietic Stem Cells in Transfusion-dependent β Thalassemia Patients
Brief Title: Safety and Efficacy Evaluation of Autologous CRISPR-Cas12b Edited Hematopoietic Stem Cells
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Shanghai Vitalgen BioPharma Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Shi, Director of Regenerative Medical Center, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGB-Ex01-001
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Thalassemia, Beta; Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VGB-Ex01 (Experimental): Each subject will accept one dose of VGB-Ex01.
  Interventions: Biological: VGB-Ex01

INTERVENTIONS:
Biological: VGB-Ex01 — CRISPR-Cas12b editing hematopoietic stem cells

SUMMARY:
This is a single-arm, open, single-injection exploratory clinical study with two transfusion-dependent β thalassemia (β-TDT) participants planned to enroll.

DETAILED DESCRIPTION:
Through CRISPR-Cas 12b editing tool with independent intellectual property rights of Chinese Academy of Sciences, HBG1/2 promoter was edited to reactivate gamma-globin and induce fetal hemoglobin (HbF) expression. This leads to a subsequent reduction in ineffective red blood cell production (due to a reduction in the uncompounded alpha-globin chain) and improved red blood cell survival (due to reduced hemolysis), ultimately improving the sequelae of anemia and reducing the need for transfusion. Safety and efficacy will be evaluated continuously throughout the study, follow-up was up to 24 months. After the end of this trial, participants who received the infusion of autologous CRISPR-Cas12b edited hematopoietic stem cells (VGB-Ex01) will be invited to participate in the long-term follow-up study to complete the 15-year follow-up plan.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-35 years old (inclusive), male or female;
* The subject and/or his/her legally recognized representative/parent/guardian fully understands the study and all information related to the study and has signed the informed consent form;
* Clinical diagnosis of transfusion-dependent β-thalassemia (TDT) with a blood transfusion record within 2 years (inclusive) prior to screening showing a history of ≥ 10 units (U)/kg/year (or ≥ 100 mL/kg/year) or ≥ 8 times/year of suspended RBC transfusions in at least 1 consecutive 12-month period;
* Karnofsky score (for subjects aged ≥ 16 years) or Lansky score (for subjects aged < 16 years) of ≥ 80;
* Subjects in stable disease state who are eligible for hematopoietic stem cell transplantation as per investigator's judgment;
* Access to diagnosis and treatment records issued by medical professional institutions within 2 years prior to screening, including the records of blood transfusions, hematology, serum chemistry, and other examinations;
* Willing and able to comply with study procedures, with good compliance, and willing to receive and complete the follow-up study with a duration of at least 2 years;
* Subjects of childbearing potential (including female subjects of childbearing potential and male subjects whose partners are of childbearing potential) must use effective contraception within 12 months of treatment.

Exclusion Criteria:

* Diagnosis of associated α-thalassemia: > 1 alpha chain deletion or alpha gene functional defect;
* Have available HLA-fully matched donors and acceptable for allogeneic hematopoietic stem cell transplantation;
* Irregular antibody or platelet antibody positive;
* Prior allogeneic bone marrow transplantation or gene therapy;
* Subjects with clinically significant and active bacterial, viral, fungal, or parasitic infection as determined by the investigator at screening, including but not limited to those with positive etiology of human immunodeficiency virus (HIV-1/2), human cytomegalovirus (HCMV-DNA), Epstein-Barr virus (EBV-DNA), or Treponema pallidum antibody (TP-Ab), or with previous hepatitis B or C infection;
* Subjects with an injury of major organs
* Contraindications for hematopoietic stem cell collection and poor collection efficiency judged by the investigator;
* Contraindications to the clinical investigational product and its excipients, G-CSF (hematopoietic stem cell mobilization), plerixafor (hematopoietic stem cell mobilization), busulfan (myeloablation), and other drugs;
* Participation within 3 months prior to screening or current participation in another interventional clinical study;
* History or family history of malignancy or myeloproliferative disorder;
* History of uncontrollable epilepsy, mental disorder, or other psychiatric disorders;
* Abuse of psychoactive substance, drug, or alcohol within 6 months prior to enrollment;
* Pregnant or breastfeeding females;
* Other diseases or reasons that interfere with study procedures;
* Any other conditions that the investigator deems unsuitable for the subject's participation in the study.

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events | Baseline up to 24 months
  An adverse event is any untoward medical occurrence in a clinical investigation/participant administered a product; the event will not need to have a causal relationship with the treatment. A serious adverse event is any untoward medical occurrence at any dose that resulted in death; life threatening;require inpatient hospitalization or prolongation of existing hospitalization; result in persistent or significant disability/incapacity; result in congenital anomaly/birth defect.
Number of subjects with neutrophil implantation ≤ 42 days | Baseline up to 42 days
  Neutrophil implantation was defined as 3 consecutive days with 3 tests for ANC≥500/μL.

SECONDARY OUTCOMES:
Number of subjects transfusion independence (TI) for at least 6 months after transfusion | Baseline up to 6 months
  TI defined as Hb≥9g/dL without red blood cell infusion
Number of subjects transfusion independence (TI) for at least 12 months after transfusion | Baseline up to 12 months
  TI defined as Hb≥9g/dL without red blood cell infusion
Fetal hemoglobin (HbF) concentration | Baseline up to 24 months
  Changes in HbF concentration from baseline after transfusion
Total hemoglobin (Hb) concentration | Baseline up to 24 months
  Changes in Hb concentration compared with baseline after transfusion
The proportion of circulating red blood cells | Baseline up to 24 months
  Changes in the proportion of circulating red blood cells expressing fetal hemoglobin compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jun Shi, PhD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Regenerative Medicine Center, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No